CLINICAL TRIAL: NCT02829138
Title: Personalized Nutrition in Young Adults: The Ability of Genetic Information to Motivate Changes in Omega-3 Consumption
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Guelph (Other)
Responsible Party: Principal Investigator, David M Mutch, Dr. David Mutch, PhD, University of Guelph
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: Personalized Nutrition
Record Dates: First submitted 2016-07-06; First posted 2016-07-12 (Estimated); Results first posted 2018-01-09 (Actual); Last update posted 2018-02-05 (Actual); Status verified 2018-01

CONDITIONS: Health Behaviour; Nutrition Intervention; Impaired Health

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Non-genetic Group (Placebo Comparator): General Nutrition related to Omega-3 fats: Individuals in this group will be provided with only general nutrition information related to omega-3 fats and health.
  Interventions: Behavioral: General Nutrition related to Omega-3 fats
- Genetic Group (Experimental): Genetic information and Omega-3 fat intake: Individuals in this group will be provided with general nutrition information related to omega-3 fats and health, as well as their personal genetic information for a common gene variant related to omega-3 fatty acid metabolism.
  Interventions: Genetic: Genetic information and Omega-3 fat intake; Behavioral: General Nutrition related to Omega-3 fats

INTERVENTIONS:
Genetic: Genetic information and Omega-3 fat intake — Only the Genetic group will receive their personal genetic information prior to beginning the 3-month study.
  Arms: Genetic Group
Behavioral: General Nutrition related to Omega-3 fats — Both the Genetic and Non-Genetic groups will receive general nutrition information about omega-3 fats.

SUMMARY:
There are many health benefits associated with the consumption of omega-3 dietary fats. Omega-3 fats, specifically eicosapentaenoic acid (EPA) and docosahexaenoic acid (DHA), can be found in marine food products such as fatty fish, in fortified products such as eggs and milk, or in dietary supplements such as fish oil. Despite numerous health benefits, it is well documented that most people in Western society are not meeting the recommended daily amounts of EPA and DHA omega-3 fats.

The overall objective of this study is to examine whether providing young adults (18-25 years) with personal genetic information changes behavior with regards to omega-3 fat consumption. In order to achieve this objective, study participants will be divided into two groups: 1. Genetic and 2. Non-Genetic. The Genetic Group will be provided with their personalized information regarding a common gene variant in addition to general information regarding the health benefits of omega-3 fats, while the Non-Genetic Group will only receive the general information. Primary outcomes studied will include dietary habits and secondary outcomes include blood markers of cardiometabolic health.

DETAILED DESCRIPTION:
There are many health benefits associated with the consumption of omega-3 dietary fats. Omega-3 fats, specifically eicosapentaenoic acid (EPA) and docosahexaenoic acid (DHA), can be found in marine food products such as fatty fish, in fortified products such as eggs and milk, or in dietary supplements such as fish oil. Despite numerous health benefits, it is well documented that most people in Western society are not meeting the recommended daily amounts of EPA and DHA omega-3 fats.

The numerous health benefits associated with omega-3 fats are well documented in scientific literature; however, there are a limited number of studies focused on the health effects of omega-3 fats in emerging adults (18-25 years). Indeed, most research to date has been conducted in older adults, with or without hyperlipidemia. In addition, it is important to consider interventions in emerging adults given that behaviours learned in this life stage can persist later in life. It has also been reported that the diet quality (i.e., amount of fruits, vegetables, whole grains, etc.) is reduced for individuals within this age range; thus highlighting another important reason for targeting this demographic.

The combination of genetic and dietary information (i.e., nutrigenetics) has the potential to not only benefit basic research, but also the general population. Therefore, more research is needed to determine if providing individuals with their genetic information has the potential to encourage behaviour changes. So far, several studies have investigated how people may change their behaviour in response to genetic risk information, but none have conducted a nutrigenetic intervention examining if providing personal genetic information alters diet behaviours.

The overall objective of this study is to examine whether providing emerging adults with personal genetic information changes their behavior with regards to omega-3 consumption. In order to achieve this objective, study participants will be divided into two groups: 1. Genetic and 2. Non-genetic. The Genetic group will be provided with their personal information for a common gene variant in addition to general information regarding the health benefits of omega-3 fats, while the Non-genetic group will only receive the general information. Primary outcomes studied will include dietary habits and secondary outcomes include blood markers of cardiometabolic health.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18-25 years

Exclusion Criteria:

* Younger than 18 years
* Older than 25 years
* Allergic to fish and/or shellfish
* If the participants are currently consuming high amounts of omega-3 food products
* Unable to get to the University of Guelph for study visits (lack of transportation, or lives too far away)
* Anticipating a significant change in lifestyle (moving houses, joining the gym, participating in elite athletic activities)
* Not comfortable giving blood samples
* Taking medication which modifies or changes blood lipid levels
* Expecting to become pregnant, pregnant or lactating

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 57 (Actual)
Dates: Start 2015-08; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David M Mutch, PhD, Principal Investigator — University of Guelph

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tur JA, Bibiloni MM, Sureda A, Pons A. Dietary sources of omega 3 fatty acids: public health risks and benefits. Br J Nutr. 2012 Jun;107 Suppl 2:S23-52. doi: 10.1017/S0007114512001456. PMID 22591897
- [Background] Micha R, Khatibzadeh S, Shi P, Fahimi S, Lim S, Andrews KG, Engell RE, Powles J, Ezzati M, Mozaffarian D; Global Burden of Diseases Nutrition and Chronic Diseases Expert Group NutriCoDE. Global, regional, and national consumption levels of dietary fats and oils in 1990 and 2010: a systematic analysis including 266 country-specific nutrition surveys. BMJ. 2014 Apr 15;348:g2272. doi: 10.1136/bmj.g2272. PMID 24736206
- [Background] Beasley LJ, Hackett AF, Maxwell SM. The dietary and health behaviour of young people aged 18-25 years living independently or in the family home in Liverpool, UK. International Journal of Consumer Studies 28(4): 355-363, 2004.
- [Background] Demory-Luce D, Morales M, Nicklas T, Baranowski T, Zakeri I, Berenson G. Changes in food group consumption patterns from childhood to young adulthood: the Bogalusa Heart Study. J Am Diet Assoc. 2004 Nov;104(11):1684-91. doi: 10.1016/j.jada.2004.07.026. PMID 15499355
- [Background] McBride CM, Koehly LM, Sanderson SC, Kaphingst KA. The behavioral response to personalized genetic information: will genetic risk profiles motivate individuals and families to choose more healthful behaviors? Annu Rev Public Health. 2010;31:89-103. doi: 10.1146/annurev.publhealth.012809.103532. PMID 20070198
- [Result] Roke K, Walton K, Klingel SL, Harnett A, Subedi S, Haines J, Mutch DM. Evaluating Changes in Omega-3 Fatty Acid Intake after Receiving Personal FADS1 Genetic Information: A Randomized Nutrigenetic Intervention. Nutrients. 2017 Mar 6;9(3):240. doi: 10.3390/nu9030240. PMID 28272299

RESULTS

PARTICIPANT FLOW:
Groups:
- Non-genetic Group: General Nutrition related to Omega-3 fats: Individuals in this group were provided with only general nutrition information related to omega-3 fats and health.
- Genetic Group: Genetic information and Omega-3 fat intake: Individuals in this group were provided with general nutrition information related to omega-3 fats and health, as well as information regarding the impact of a common variant in the FADS1 gene and how this variant influences omega-3 fatty acid profiles.
Period: Overall Study
Arm/Group | Non-genetic Group | Genetic Group
Started | 29 | 28
Completed | 28 | 28
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Non-genetic Group | Genetic Group | Total
Number analyzed (Participants) | 29 | 28 | 57
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 29 | 28 | 57
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 28 | 57
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Canada | 29 | 28 | 57

OUTCOME MEASURES:

1. Primary Outcome: Omega-3 Dietary Intake
Description: Omega-3 fat intake was assessed using food frequency questionnaires. The Canadian Nutrient File (version 2015) was used to assess the amount of EPA and DHA in whole foods (e.g., fish, eggs, poultry). Data corresponds to EPA + DHA (mg /day).
Time Frame: Baseline and 12 weeks
Measure: Mean (Standard Error); unit: mg/day
Arm/Group | Non-genetic Group | Genetic Group
Number analyzed (Participants) | 28 | 28
mg/day
  Baseline | 190.16 (39.21) | 211.50 (43.16)
  12 weeks | 395.82 (70.60) | 323.23 (65.27)

2. Secondary Outcome: Change in Blood Triglycerides (Physiological Parameter)
Description: Triglycerides were measured in fasted serum. Data is reported as mmol/L
Time Frame: baseline and 12 weeks
Measure: Mean (Standard Error); unit: mmol/L
Arm/Group | Non-genetic Group | Genetic Group
Number analyzed (Participants) | 28 | 28
mmol/L
  Baseline | 1.02 (0.07) | 0.9 (0.07)
  12 weeks | 1.02 (0.06) | 1.02 (0.08)

3. Secondary Outcome: Change in Omega-3 Index in Blood (Physiological Parameter)
Description: Blood fatty acids measured by gas chromatography. Data is reported as a percentage of all detected fatty acids. The omega-3 index is calculated by summing data for 3 omega-3 fats in serum: ALA, EPA, and DHA.
Time Frame: baseline and 12 weeks
Measure: Mean (Standard Error); unit: percentage of total fatty acids in serum
Arm/Group | Non-genetic Group | Genetic Group
Number analyzed (Participants) | 28 | 28
percentage of total fatty acids in serum
  Baseline | 3.97 (0.12) | 3.86 (0.11)
  12 weeks | 4.15 (0.13) | 3.97 (0.11)

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Non-genetic Group | Genetic Group
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/28
Other Adverse Events (participants affected / at risk) | 0/28 | 0/28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No